CLINICAL TRIAL: NCT01053676
Title: Bioequivalence Study of BAY77-1931 Granule - Randomized, Non-blind, Two-way, Crossover Study to Establish the Bioequivalence Between BAY77-1931 Granule 500 mg and Fosrenol Chewable Tablet 500 mg in Japanese Healthy Male Adult Subjects
Brief Title: Bioequivalence Study of BAY77-1931 Granule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13287
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Hyperphosphatemia
Keywords: Hyperphosphatemia; BE; Granule; Healthy volunteers
MeSH Terms: conditions — Hyperphosphatemia | interventions — lanthanum carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Lanthanum Carbonate (Fosrenol, BAY77-1931) Granule
- Arm 2 (Active Comparator)
  Interventions: Drug: Lanthanum Carbonate (Fosrenol, BAY77-1931) Chewable tablet

INTERVENTIONS:
Drug: Lanthanum Carbonate (Fosrenol, BAY77-1931) Granule — BAY77-1931 Granule TID for 4 days
  Arms: Arm 1
Drug: Lanthanum Carbonate (Fosrenol, BAY77-1931) Chewable tablet — BAY77-1931 Chewable tablet TID for 4 days
  Arms: Arm 2

SUMMARY:
The study is conducted as a randomized, non-blinded, 2-way crossover study. Target population is 60 Japanese healthy male adult subjects selected by screening examination which will be conducted within 4 weeks before the first drug administration of period 1 (before the hospitalization of period 1). Subjects will admit in the clinical institute on Day -3 and be discharged on Day 6 in each period. During hospitalization, standardized phosphate diet from Day -2 to Day 4 will start approximately 20 minutes before dosing. Subject will take about 1300 mg of phosphate evenly at breakfast lunch and dinner for each day. Subject should consume at least 95% of a meal. Distilled water not to include phosphate will be used for drinking water and meal. Subjects are to drink at least 1 L of distilled water every day in clinic to make sure enough urine volume. The 24 hours urine collection will be conducted between Day -2 and Day 4 to investigate the urinary phosphate excretion.BAY77-1931 granule 500 mg or Fosrenol chewable tablet 500 mg will be administered three times daily after each meal from Day 1 to Day 4. On day 4 single dose after breakfast will be administered. Study drugs will be administered immediately after each meal, that is within 20 minutes after start of each meal with 240 mL of distilled water. A Fosrenol chewable tablet 500 mg will be taken after chewing completely.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male volunteers who must have given their written informed consent to participate in the study
* Age is between 20 and 45 years
* Body Mass Index (BMI) is between 17.6 and 26.4 kg/m2.
* Volunteers who are judged by the investigators to be suitable for enrollment in this clinical trial based upon the data from a screening test.

Exclusion Criteria:

* A history of relevant diseases of internal organs (diseases that may significantly jeopardize body systems, such as severe liver or renal dysfunction, active peptic ulcer, ulcerative colitis, Crohn's disease, narrowing of colon lumen) or, of the central nervous system (e.g., epilepsy), or other organs which are likely to show inappropriateness for participation in this study
* Conditions of such that would impair the subject's ability to participate or complete this study in the opinion of the investigator (mental diseases that are thought to be ineligible for the communal life in the study participation, unable to consent to the participation, disables)
* Known drug hypersensitivity or idiosyncrasy

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on daily urinary phosphate excretion | Follow up examination cunducted on 7 to 10 days after the last drug administration

SECONDARY OUTCOMES:
Adverse event collection | Follow up examination cunducted on 7 to 10 days after the last drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Osaka, Osaka, Japan